CLINICAL TRIAL: NCT04658550
Title: A Mixed Retrospective-prospective, Observational Study Evaluating the Efficacy of Counselling in a Remote Setting Compared to an In-person Setting on Weight Loss, in Obese Patients With Body Mass Index > 35 Kg/m2 and Enrolled in the Behaviour Modification Program at the Bariatric Centre of Excellence at St Joseph's Healthcare Hamilton.
Brief Title: Remote vs In Person Weight Loss Study
Status: Completed | Type: Observational
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Tony Chetty, Associate Professor Pathology and Molecular Medicine, St. Joseph's Healthcare Hamilton
Other Study IDs: Remote v In Person Weight Loss
Record Dates: First submitted 2020-10-09; First posted 2020-12-08 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Remote Weight Loss Behaviour Modification Program with Meal Replacements: This is the prospective study group who will receive 26-weeks of weight loss and maintenance counselling in a remote setting and a low-calorie meal replacement as part of their usual care.
  Interventions: Other: Remote Behaviour Modification Program
- In Person Weight Bahaviour Modification Program with Meal Replacements: This is the retrospective study group who received 26-weeks of weight loss and maintenance counselling in person and a low-calorie meal replacement as part of their usual care.
  Interventions: Other: In Person Behaviour Modification Program

INTERVENTIONS:
Other: Remote Behaviour Modification Program — The standard of care behaviour modification program for weight loss will be offered virtually due to the COVID-19 pandemic (prospective).
  Groups: Remote Weight Loss Behaviour Modification Program with Meal Replacements
Other: In Person Behaviour Modification Program — The standard of care behaviour modification program for weight loss was offered in person prior to the COVID-19 pandemic (retrospective).
  Groups: In Person Weight Bahaviour Modification Program with Meal Replacements

SUMMARY:
The COVID-19 pandemic has created fear, financial difficulties and interruptions in the lives of patients and healthcare providers. As a result, many patients suffering from chronic conditions such as obesity have had their treatment disrupted by the pandemic. The Bariatric Medical Weight Management Clinic at St. Joseph's Healthcare Hamilton transitioned its weight loss and maintenance counselling classes to a remote (online) platform in response to the pandemic. The remote weight loss and maintenance classes allows patients to continue receiving treatment for obesity from their homes. The remote weight loss and maintenance program is conducted on a safe platform that has been thoroughly reviewed and approved by St. Joseph's Privacy Committees.

The aim of this study is to learn whether the remote weight loss and maintenance classes can lead to similar weight loss compared to the in-person weight loss and maintenance classes that were offered to patients before the COVID-19 pandemic. This study also aims to gather feedback about the program to improve its delivery and patients' experiences.

DETAILED DESCRIPTION:
The COVID-19 pandemic has created fear, financial difficulties and interruptions in the lives of patients and healthcare providers. As a result, many patients suffering from chronic conditions such as obesity have had their treatment disrupted by the pandemic. The Bariatric Medical Weight Management Clinic at St. Joseph's Healthcare Hamilton transitioned its behaviour modification program, also known as weight loss and maintenance counselling classes, to a remote (online) platform in response to the pandemic. The remote weight loss and maintenance classes allow patients to continue receiving treatment for obesity from their homes.

This is a 26-week, single-centre, mixed retrospective and prospective, observational study evaluating the efficacy of counselling in a remote setting compared to an in-person setting in achieving weight loss among adult patients with obesity enrolled in the behaviour modification program. This study also aims to gather feedback about the program to improve its delivery and patients' experiences.

Approximately 120 patients participating in the behaviour modification program and providing informed consent will be observed in this study. This study involves a prospective and retrospective component. The prospective component will be an observational study of 60 subjects who will receive 26-weeks of weight loss and maintenance counselling in a remote setting and a low-calorie meal replacement as part of their usual care. The retrospective component will involve using historical data from 60 subjects who received 26-weeks of weight loss and maintenance counselling in an in-person setting and a low-calorie meal replacement as part of their usual care.

Parameters measured as part of standard of care at the start and end of the program, such as body weight, blood pressure and lab tests will be collected for analysis of study endpoints. Participants will also be asked to complete a satisfaction survey at the end. There will be no blinding of patients, study investigators, or data analysts.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Enrolled in 26-week BCoE behaviour modification program with meal replacements
* Able and willing to provide signed informed consent

Exclusion Criteria:

- Subjects will be excluded if they contact clinic or study personnel to withdraw consent or withdraw data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients with Body Mass Index > 35 Kg/m2 and enrolled in the behaviour modification program for weight loss at the Bariatric Centre of Excellence at St Joseph's Healthcare Hamilton
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mean Percentage Change in Body Weight | Baseline to Week 26
  To evaluate the efficacy of counselling in a remote setting compared to an in-person setting in achieving weight loss among adult patients with obesity enrolled in the behaviour modification program

SECONDARY OUTCOMES:
Patient satisfaction and barriers to participation | Week 26
  Patient satisfaction and barriers to participation associated with the remote weight loss and maintenance program as assessed by the Bariatric Centre of Excellence Virtual Medical Program Satisfaction Survey.
Change in blood pressure | Baseline to Week 26
  Change in blood pressure
Change in lipid profile | Baseline to Week 26
  Change in lipid profile including total cholesterol, triglycerides, low density lipoprotein and high density lipoprotein
Change in fasting blood glucose | Baseline to Week 26
  Change in fasting blood glucose
Change in heart rate | Baseline to Week 26
  Change in heart rate
Change in HbA1C | Baseline to Week 26
  Change in HbA1C

CONTACTS AND LOCATIONS:
Overall Officials: Tony Chetty, MD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No